CLINICAL TRIAL: NCT03775525
Title: A Phase I/Ib, Multicenter, Open-label, Dose-Escalation, Safety, Pharmacodynamic and Pharmacokinetic Study of GZ17-6.02 Monotherapy and in Combination With Capecitabine, Given Orally on a Daily Schedule in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Study Evaluating GZ17-6.02 in Patients With Advanced Solid Tumors or in Combination With Capecitabine in Metastatic Hormone Receptor Positive Breast Cancer
Acronym: GEN602
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genzada Pharmaceuticals USA, Inc. (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEN-602-CT-101
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Advanced Cancer; Gastric Cancer; Breast Cancer; Pancreatic Cancer; Prostate Cancer Metastatic; Colo-rectal Cancer; Solid Tumor; Solid Carcinoma; Solid Carcinoma of Stomach; Cancer of Stomach; Lymphoma; Sarcoma; Cutaneous T Cell Lymphoma; Head and Neck Squamous Cell Carcinoma; Basal Cell Carcinoma; Cutaneous T-cell Lymphoma; Cutaneous Squamous Cell Carcinoma
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Lymphoma; Sarcoma; Lymphoma, T-Cell, Cutaneous; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Basal Cell | interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: monotherapy (Experimental): GZ17-6.02 given orally on a daily x 28 day schedule. This will be a dose escalation study.
  Interventions: Drug: GZ17-6.02
- Experimental: Combination with Capecitabine in Metastatic Hormone Receptor Positive Breast Cancer (Experimental): GZ17-6.02 given orally twice daily x 21 day schedule in combination with Capecitabine 825 mg/m2 orally twice daily for 14 days x 21 day schedule.
  Interventions: Drug: GZ17-6.02; Drug: Capecitabine
- Experimental: Combination with Capecitabine in Metastatic Colorectal Cancer (Experimental): GZ17-6.02 given orally twice daily x 21 day schedule in combination with Capecitabine 850 mg/m2 orally twice daily for 14 days x 21 day schedule.
  Interventions: Drug: GZ17-6.02; Drug: Capecitabine

INTERVENTIONS:
Drug: GZ17-6.02 — Super enhancer Inhibition
Drug: Capecitabine — antimetabolite
  Other Names: Xeloda
  Arms: Experimental: Combination with Capecitabine in Metastatic Colorectal Cancer; Experimental: Combination with Capecitabine in Metastatic Hormone Receptor Positive Breast Cancer

SUMMARY:
This Phase I/Ib study is a Multicenter, Open-label, Dose-Escalation, Safety, Pharmacodynamic and Pharmacokinetic Study of GZ17-6.02 Monotherapy and in Combination with Capecitabine, Given Orally on a Daily Schedule in Patients with Advanced Solid Tumors or Lymphoma

DETAILED DESCRIPTION:
This study will evaluate the safety, pharmacokinetics, and pharmacodynamic effects of a novel anti-cancer drug, GZ17-6.02 administered to patients with advanced solid tumors or lymphoma, which have progressed after receiving standard/approved therapy or where there is no approved therapy.

This study will determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of GZ17-6.02 monotherapy and in combination with standard-of-care oncology treatments and to establish the dose of GZ17-6.02 recommended for future monotherapy and combination therapies phase II oncology clinical studies.

ELIGIBILITY:
General Inclusion Criteria:

* Patients with a pathologically confirmed diagnosis of advanced solid tumors or lymphoma.
* Tumor progression after receiving standard/approved therapies which may include chemotherapy, targeted agents, radio-immuno conjugates, check point inhibitors, where there is no approved therapy; or the patient is intolerant of standard of care or the patient declines standard of care treatment
* One or more metastatic tumors measurable, or evaluable, per RECIST v1.1 Criteria for solid tumors and Lugano Criteria for lymphoma
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Life expectancy of at least 3 months
* Age 18 years
* Signed, written IRB-approved informed consent
* A negative pregnancy test (if female)
* Acceptable liver function:

  * Bilirubin ≤ 1.5 times upper limit of normal
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase ≤ 2.5 times upper limit of normal (if liver metastases are present, then ≤ 5 x ULN is allowed)
* Acceptable renal function:

  o Serum creatinine ≤ 1.5 times institutional ULN, OR calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Acceptable hematologic status:

  * Granulocyte ≥ 1500 cells/mm3
  * Platelet count ≥ 100,000 (plt/mm3)
  * Hemoglobin ≥ 9 g/dL
* Urinalysis:

  o No clinically significant abnormalities
* Acceptable coagulation status (for patients on warfarin or other anti-coagulants, a PT/PTT considered by the PI as therapeutically appropriate will be allowed):

  * PT within ≤ 1.5 times normal limits
  * PTT within ≤ 1.5 times normal limits
* For men and women of child-producing potential, the use of effective contraceptive methods during the study
* Fasting glucose ≤ 180 mg/dL
* Albumin ≥ 3.0 g/dL within seven days of initiating protocol treatment

For patients in the GZ17-6.02 plus capecitabine Phase 1b Expansion Cohort 2 (metastatic breast cancer):

* Pathologically confirmed diagnosis of HER2-negative and Hormone Receptor (HR) (estrogen receptor [ER] and/or progesterone receptor)-positive metastatic breast cancer;
* Had ≤ 1 prior treatment (not including neoadjuvant or adjuvant treatment);
* Are naïve to capecitabine but not necessarily to fluorouracil (5 FU);
* Eligible for standard-of-care treatment with capecitabine monotherapy.
* Patients in Expansion Cohort 2 with bone-only metastatic disease must have one or more lytic or a mixed lytic-blastic lesions that can be assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI).

For patients in GZ17-6.02 plus capecitabine Phase 1b Expansion Cohort 3 (metastatic colorectal cancer):

* Pathologically confirmed diagnosis of metastatic colorectal cancer;
* Had ≤ 2 prior treatments (not including neoadjuvant or adjuvant treatment);
* Are naïve to capecitabine but not necessarily to 5 FU;
* Eligible for standard-of-care treatment with capecitabine monotherapy.

General Exclusion Criteria: (All patients, unless otherwise specified):

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG.
* Currently taking MAOIs
* Baseline QTc exceeding 450 msec in males, 470 msec in females (using the Fridericia's formula) and/or patients receiving class 1A or class III antiarrhythmic agents;
* Known active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy;
* Pregnant or nursing women.
* NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Treatment with radiation therapy or surgery within 1 month prior to study entry.
* Treatment with chemotherapy, targeted therapeutics (e.g. tyrosine kinase inhibitors, therapeutic antibodies, etc), or investigational therapies within 1 month, or 5 half-lives (whichever is shorter), prior to study entry (6 weeks for nitrosoureas or mitomycin C). For radiopharmaceuticals, within 1 month unless hematopoietic recovery has not returned to pretreatment baseline;
* Unwillingness or inability to comply with procedures required in this protocol;
* Known active infection with HIV, HTLV-1, hepatitis B, hepatitis C or other chronic viral infections that could interfere with the interpretation of study data;
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor.
* Patients who are currently receiving any other investigational agent;
* Primary Central Nervous System (CNS) malignancies;
* Active CNS metastases requiring treatment or radiotherapy, or which have not been confirmed stable on radiographic imaging for ≥30 days prior to C1D1;
* Patients requiring steroids for neurological signs and symptom stabilization.
* Patients who are unable to successfully discontinue all prohibited medications listed in Appendix 6;
* Patients must not have received a transfusion (platelets or red blood cells) ≤ 2 weeks prior to initiating protocol therapy.

For patients in the GZ17-6.02 monotherapy Dose Escalation Cohort and patients in Expansion Cohort 1:

• Patients with cow's milk allergy or with galactosemia

Phase 1b Expansion Cohort 2 (metastatic breast cancer) and Expansion Cohort 3 (metastatic colorectal cancer):

* Any history of coronary artery disease is exclusionary; New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on the ECG.
* Any conditions or medications that are contraindicated with capecitabine dosing;
* Dihydropyrimidine dehydrogenase (DPD) deficiency;
* Known sensitivity to capecitabine or any of its components or to 5-FU ;
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor

  o This includes prior gastrointestinal surgery that would interfere with the oral drug absorption.
* Malignancy other than metastatic breast cancer (Expansion Cohort 2) or metastatic colorectal cancer (Expansion Cohort 3) that required therapy within the preceding 5 years, other than adequately treated:

  * non-melanoma skin cancer or in situ cancer;
  * another cancer that has a very low risk of interfering with the safety or efficacy endpoints of the study, must be approved by the Sponsor medical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 18 months
  As assessed by CTCAE v4.03
Recommended dose of GZ17-6.02 for future phase II clinical studies | 18 months
Dose-limiting toxicity | 18 months

SECONDARY OUTCOMES:
Antitumor effect | 18 months
Area Under Concentration Curve | 18 months
Maximum Plasma Concentration (Cmax) | 18 months
Time to Maximum Plasma Concentration (Tmax) | 18 months
Terminal Phase Half-Life (t1/2) | 18 months
Total Body Clearance (CL/F) | 18 months
Apparent Volume of Distribution (Vd/F) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Gazarik, Study Director — Translational Drug Development
Locations (4):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth L, West C, Von Hoff D, Dent P. Mechanisms of GZ17-6.02 resistance. Anticancer Drugs. 2022 Jun 1;33(5):415-423. doi: 10.1097/CAD.0000000000001203. PMID 35276694